## **Study Information Sheet for Clinicians**

Study Title: A pilot study to test the acceptability and feasibility of a brief discussion to help patients formulate their goals for medical care in the emergency department

Version: 5/24/2017

Principal Investigator (PI): Kei Ouchi, MD, MPH

NCT03208530

**Study Information Sheet for ED Clinicians** 

Study Title: A pilot study to test the acceptability and feasibility of brief motivational interview

intervention to help patients formulate their goals for medical care in the emergency department

Principal Investigator: Kei Ouchi, MD, MPH

Purpose of the Research: This is a research study to test the acceptability and feasibility of

our brief motivational interview intervention to facilitate advance care planning (ACP)

conversation on older adults with serious co-morbid illness being discharged from the

emergency department (ED).

**Sponsor of the Research:** Emergency Medicine Foundation.

How we obtained your name and contact information: The participants are identified based

on their clinical roles as attending physicians and physician assistants belonging to the

Department of Emergency Medicine at Brigham and Women's Hospital. We inquired your

directors of service to identify you.

Why are we asking you to participate?

We are asking you to participate because we want to test the acceptability of our intervention

when performed in the ED.

How many people are anticipated to participate?

We hope to recruit 5 to 10 attending physicians and 5 to 10 physician assistants to participate in

this study.

How long it will take to complete the study?

The study will take place in the ED observation unit. We anticipate that each patient

encounter/intervention administration and answering of acceptability survey will add 8 minutes

total to you routine clinical practice. We will plan to continue enrollment until we complete 100

patient encounters total.

**Remuneration:** There is no remuneration for this study.

**Confidentiality and Data Security** 

The data will be collected in the form of qualitative (e.g. your comments) and quantitative (e.g.

how many minutes does it take to read off the scripted text in a simulated patient encounter

settings) formats. All data will be de-identified (we will not be able to match specific data to specific participant) and stored in a secure location in PI's office, which will be destroyed upon completion of the intervention development.

## What are the risks associated with participation?

There is no clear foreseeable risk associated with participation in this study other than 8 extra minutes of your time during your routine clinical practice in the ED observation unit. Your participation is voluntary and you may stop at any time.

## Questions:

The PI can be contacted at the following 24 hours / day and 7 days per week:

Cell – 857-205-4947

Email - kouchi@partners.org

If you'd like to speak to someone not involved in this research about your rights as a research subject, or any concerns or complaints you may have about the research, contact the Partners Human Research Committee at 617-424-4100.